CLINICAL TRIAL: NCT02107820
Title: Does Bladder Training (BT) Improve the Efficacy of Percutaneous Tibial Nerve Stimulation (PTNS) in Women With Refractory Overactive Bladder (OAB) - A Randomised Controlled Study
Brief Title: Does Bladder Training Improve the Efficacy of Nerve Stimulation in Women With Refractory Overactive Bladders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/P/036
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Overactive Bladder
Keywords: Bladder training; Percutaneous Tibial nerve stimulation; Overactive bladder; Randomised controlled study
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous Tibial Nerve stimulation (Active Comparator): A needle electrode insertion site is located on the inner aspect of either leg approximately three fingerbreadths (5 cm or 2") cephalad to the medial malleolus and approximately one fingerbreadth (2 cm or ¾") posterior to the tibia. The needle electrode head is gently tapped to pierce the skin, maintaining a 60° angle, and insert to a depth of approximately 2cm. The electrode is then connected to the stimulator and the current setting needed is determined by the test mode on the stimulator. Once the current setting is known, the stimulator is started on the therapy mode which delivers the current for 30 minutes and shuts off automatically after 30 minutes. The needle is then removed and stimulator disconnected. The treatment involves twelve weekly sessions of 30 minutes each.
  Interventions: Device: Percutaneous Tibial Nerve stimulation
- 'Bladder Training (BT) and PTNS (Experimental): All patients randomised to PTNS + BT group will have BT with the nurse for 20 minutes during PTNS sessions (which last 30 minutes). Since BT is recommended by NICE for a duration of 6 weeks. BT will be discussed for the first 6 sessions of the 12 week PTNS treatment cycle.
  Interventions: Behavioral: Bladder Training (BT); Device: Percutaneous Tibial Nerve stimulation

INTERVENTIONS:
Behavioral: Bladder Training (BT) — All patients randomised to PTNS + BT group will have BT with the nurse for 20 minutes during PTNS sessions (which last 30 minutes). Since BT is recommended by NICE for a duration of 6 weeks. BT will be discussed for the first 6 sessions of the 12 week PTNS treatment cycle.
  Arms: 'Bladder Training (BT) and PTNS
Device: Percutaneous Tibial Nerve stimulation — A needle electrode insertion site is located on the inner aspect of either leg approximately three fingerbreadths (5 cm or 2") cephalad to the medial malleolus and approximately one fingerbreadth (2 cm or ¾") posterior to the tibia. The needle electrode head is gently tapped to pierce the skin, maintaining a 60° angle, and insert to a depth of approximately 2cm. The electrode is then connected to the stimulator and the current setting needed is determined by the test mode on the stimulator. Once the current setting is known, the stimulator is started on the therapy mode which delivers the current for 30 minutes and shuts off automatically after 30 minutes. The needle is then removed and stimulator disconnected. The treatment involves twelve weekly sessions of 30 minutes each.

SUMMARY:
Overactive Bladder (OAB) is a chronic condition defined as urgency with or without incontinence usually associated with frequency and nocturia. It is a common condition affecting 15-45% of adults and constitutes a significant proportion of patients attending urogynaecology clinics. OAB is known to have a significant impact on the physical, social and emotional quality of life and sexual function in women. The treatment of OAB is initially conservative with bladder training followed by pharmacotherapy.

Evidence from a recent Cochrane review on treatment of OAB suggests that the efficacy of anticholinergics in treatment of OAB is enhanced when combined with BT. Women who fail to improve with these initial measures are offered Intravesical Botox or neuromodulation in the form of Percutaneous Tibial Nerve Stimulation (PTNS) or Sacral Nerve Stimulation (SNS).

PTNS has also been shown to more effective than pharmacotherapy with anticholinergics. In 2010 National Institute of Clinical Excellences (NICE) issued guidance stating '"PTNS for OAB demonstrates effectiveness without major safety concerns"

We hypothesise that the outcome of PTNS will improve if the PTNS sessions are combined with bladder training (BT).

ELIGIBILITY:
Inclusion Criteria:

* All women with refractory OAB who are offered PTNS as a treatment option

Exclusion Criteria:

* Who cannot give informed consent.
* Women in whom PTNS is contraindicated. This includes women who have:

Gross leg oedema A pacemaker

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-07-24; Primary Completion 2019-03 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Primary outcome will reduction in number of urgency episodes (bladder diary) | 3 months
  All patients complete a bladder diary (A record of fluid intake, voided volumes, urgency and incontinence episodes for 3 days) prior to commencement and at 3 months.

SECONDARY OUTCOMES:
reduction in frequency | 24 months
  Bladder diary and International Consultation on Incontinence Questionnaire - OverActive Bladder (ICIQ-OAB) questionnaire
urgency incontinence episodes | 24 months
  ICIQ-OAB questionnaire
increase in mean void volume | 3 months
  Bladder diary
improvement in quality of life and urgency scores | 24 months
  ICIQ-OAB questionnaire

OTHER OUTCOMES:
Patient 4 point likert scale 0-3 (0 no effect, 1 better, 2 much better, 3 cured) | 24 months
  Patients are asked about the subjective effect of the treatment on a 4 point likert scale 0-3 (0 no effect, 1 better, 2 much better, 3 cured) during the treatment cycle
Patient global impression of improvement (PGII) (5 point likert scale) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anupreet Dua, MBBS, MRCOG, Principal Investigator — Plymouth Hospitals NHS Trust (PHNT)
Locations (1):
- Plymouth Hospitals NHS Trust (PHNT), Plymouth, Devon, United Kingdom